CLINICAL TRIAL: NCT05079659
Title: Rate , Predictors and Outcome of Chronic Migraine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Omar Abdeaziz, DOCTOR, Assiut University
Other Study IDs: chronic migraine
Record Dates: First submitted 2021-09-28; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Chronic Migraine, Headache; Chronic Migraine
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Nowadays, headache has been considered as one of the top global disabling medical conditions.1 Migraine is an important type of headache, and one of the chronic multifaceted neuro-inflammatory disorders.2 It is characterized by recurrent throbbing headache pain that typically affects one side of the head, and is often accompanied by nausea and disturbed vision. Migraine headache accounts for 1.4% of all neurological and mental disorders.2 It was reported that the estimated lifetime prevalence of migraine ranged 12%-18%.3 Chronic migraine is defined by the International Classification of Headache Disorders - ICHD-3 as having headaches for ≥ 15 days per month, for ≥ 3 months

, which ≥ 8 days/month are linked to migraine. Chronic migraine affects around 1%-4% of the population and chronic tension-type headache about 2.2%.4 Approximately 25%-50% of those affected also have medication overuse headache, which has a population prevalence of 1%.5 Chronic headache is a severely disabling long-term condition, with higher symptom ,frequency and severity than episodic headache.6

DETAILED DESCRIPTION:
Nowadays, headache has been considered as one of the top global disabling medical conditions.1 Migraine is an important type of headache, and one of the chronic multifaceted neuro-inflammatory disorders.2 It is characterized by recurrent throbbing headache pain that typically affects one side of the head, and is often accompanied by nausea and disturbed vision. Migraine headache accounts for 1.4% of all neurological and mental disorders.2 It was reported that the estimated lifetime prevalence of migraine ranged 12%-18%.3 Chronic migraine is defined by the International Classification of Headache Disorders - ICHD-3 as having headaches for ≥ 15 days per month, for ≥ 3 months

, which ≥ 8 days/month are linked to migraine. Chronic migraine affects around 1%-4% of the population and chronic tension-type headache about 2.2%.4 Approximately 25%-50% of those affected also have medication overuse headache, which has a population prevalence of 1%.5 Chronic headache is a severely disabling long-term condition, with higher symptom ,frequency and severity than episodic headache.6 Diagnostic criteria of chronic migraine according to ICHD(7)

Description:

Headache occurring on 15 or more days/month for more than 3 months, which, on at least 8 days/month, has the features of migraine headache.

Diagnostic criteria:

A. Headache (migraine-like or tension-type-like1) on ≥15 days/month for >3 months, and fulfilling criteria B and C B. Occurring in a patient who has had at least five attacks fulfilling criteria B-D for 1.1 Migraine without aura and/or criteria B and C for 1.2 Migraine with aura

C. On ≥8 days/month for >3 months, fulfilling any of the following:

1. criteria C and D for 1.1 Migraine without aura
2. criteria B and C for 1.2 Migraine with aura
3. elieved by the patient to be migraine at onset and relieved by a triptan or ergot derivative D Not better accounted for by another ICHD-3 diagnosis.

Episodic migraine (EM) is characterized by those with migraine who have 0 to 14 headache days per month, while chronic migraine (CM) is characterized by 15 or more headache days per month.

The relationship between EM and CM is complex. EM progresses to CM at the rate of 2.5% per year [8], and CM often remits to EM (2-year transition rate of 26%) [9].

Several factors have been associated with migraine chronification (predictors) ; such as age:

* Age *Sex *Presence of depression *Presence of anxiety
* sleep disorder *obesity *medication compliance *medication overuse
* coffee * low income *allodynia *other pain disordes comorbidities.

Our aims were to identify factors that predict prognosis in patients with chronic Migraine.

ELIGIBILITY:
Inclusion Criteria:

* 1- both sex 2- all age groups are included 3-history suggestive of chronic migraine 4-accept to participate in the study

Exclusion Criteria:

1-presence of neurological disease other than chronic migraine 2-presence of other chronic medical conditions 3-patients refuse to participate in the study .

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: sample size was calculated using epidemiological information statistical package version 7.
  Based on paramaters for cross sectional study;proportion of remitted migraine .26 ,acceptable margin of error 0.05 ,design effect1.95% confidence level.
  The required sample size will be 296 migrainous patient .
Sampling Method: Non-Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
To assess remission rate of chronic migraine to episodic migraine | 2 years
  by assessing cases which remit from chronic migraine to episodic migraine according to the criteria of each of them

SECONDARY OUTCOMES:
to assess potential predictors of chronic migraine | 2 years
  by assessing factors affecting remission of chronic migraine

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Noor T, Sajjad A, Asma A. Frequency, character and predisposing factor of headache among students of medical college of Karachi. J Pak Med Assoc. 2016 Feb;66(2):159-64. PMID 26819160
- [Background] van Hemert S, Breedveld AC, Rovers JM, Vermeiden JP, Witteman BJ, Smits MG, de Roos NM. Migraine associated with gastrointestinal disorders: review of the literature and clinical implications. Front Neurol. 2014 Nov 21;5:241. doi: 10.3389/fneur.2014.00241. eCollection 2014. PMID 25484876
- [Background] Semiz M, Senturk IA, Balaban H, Yagiz AK, Kavakci O. Prevalence of migraine and co-morbid psychiatric disorders among students of Cumhuriyet University. J Headache Pain. 2013 Apr 11;14(1):34. doi: 10.1186/1129-2377-14-34. PMID 23578213
- [Background] Ibrahim N, Al-Kharboush D, El-Khatib L, Al-Habib A, Asali D. Prevalence and Predictors of Anxiety and Depression among Female Medical Students in King Abdulaziz University, Jeddah, Saudi Arabia. Iran J Public Health. 2013 Jul 1;42(7):726-36. eCollection 2013. PMID 24427751
- [Background] Cousins G, Hijazze S, Van de Laar FA, Fahey T. Diagnostic accuracy of the ID Migraine: a systematic review and meta-analysis. Headache. 2011 Jul-Aug;51(7):1140-8. doi: 10.1111/j.1526-4610.2011.01916.x. Epub 2011 Jun 7. PMID 21649653
- [Background] Bigal ME, Serrano D, Buse D, Scher A, Stewart WF, Lipton RB. Acute migraine medications and evolution from episodic to chronic migraine: a longitudinal population-based study. Headache. 2008 Sep;48(8):1157-68. doi: 10.1111/j.1526-4610.2008.01217.x. PMID 18808500
- [Background] Manack A, Buse DC, Serrano D, Turkel CC, Lipton RB. Rates, predictors, and consequences of remission from chronic migraine to episodic migraine. Neurology. 2011 Feb 22;76(8):711-8. doi: 10.1212/WNL.0b013e31820d8af2. Epub 2011 Jan 26. PMID 21270413
- [Background] McKenna SP, Doward LC, Davey KM. The Development and Psychometric Properties of the MSQOL: A Migraine-Specific Quality-of-Life Instrument. Clin Drug Investig. 1998;15(5):413-23. doi: 10.2165/00044011-199815050-00006. PMID 18370497